CLINICAL TRIAL: NCT05737862
Title: Effect of Moringa Oleifera Leaf Capsul on Hemoglobin Levels in Anemia: A Pilot Study
Brief Title: Effect of Moringa Oleifera Leaf on Hemoglobin Levels in Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAGPH-202210.01
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Anemia of Pregnancy
MeSH Terms: interventions — Iron

STUDY DESIGN:
Intervention Model Description: 1 group receives capsules of powdered Moringa leaves (active comparator), and the other group receives IFA tablets as part of routine clinical care.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa oleifera leaf capsule (Experimental): Subjects in this arm receive experimental capsules containing powdered Moringa oleifera leaf capsules along with IFA tablets
  Interventions: Dietary Supplement: Moringa oleifera capsules; Dietary Supplement: iron and folic acid supplements
- Iron and folic acid capsule (Active Comparator): Subjects in this arm only receive iron and folic acid (IFA) tablets
  Interventions: Dietary Supplement: iron and folic acid supplements

INTERVENTIONS:
Dietary Supplement: Moringa oleifera capsules — In this arm, pregnant mothers receive capsules containing 500 mg of powdered Moringa oleifera leaves which contain 13.09 mg of iron per100 gram. Dose: 2 × 2 capsules per day for 30 days
  Arms: Moringa oleifera leaf capsule
Dietary Supplement: iron and folic acid supplements — In this arm, pregnant mothers receive IFA tablets 2 × 1 tablet a day for 30 days. Each IFA tablet contains 400 mcg folic acid and 180 mg Ferrous Fumarate.

SUMMARY:
The main objective of this study was to compare the results of hemoglobin levels between pregnant women in the treatment group and the control group. Participants will be subjected to anthropometric measurements, recall of food intake for 1 x 24 hours, check hemoglobin before and after being given the intervention and participants in the treatment group are given moringa leaf capsules and iron tablets while participants in the control group are only given iron tablets. Researchers will compare the final results of hemoglobin levels between the treatment group and the control group

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with 2nd and 3rd trimester of pregnancy
* Pregnant women with mild to moderate anemia At day 90 after treatment

Exclusion Criteria :

* Hypotensive pregnant women
* Pregnant women with Gemelli
* Pregnant women with chronic diseases (hepatitis and HIV)

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Haemoglobin (Hb) level | Day 0 and day 30
  Hb will be meassured twice, before treatment and 30 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Padjajaran, Bandung, West Java, Indonesia

DOCUMENTS (1):
  • Study Protocol (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT05737862/Prot_000.pdf